CLINICAL TRIAL: NCT00492609
Title: Medical and Economical Evaluation of Computer-assisted Reconstruction of the ACL
Brief Title: Medical and Economical Evaluation of Computer-assisted Reconstruction of the Anterior Cruciate Ligament (ACL)
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Dr Plaweski, Grenoble University Hospital
Other Study IDs: DCIC 05 47; PRAXIM SOCIETY
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament; Arthroscopy
Keywords: Surgery; Navigation; ACL; IKDC; comparative study
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: PATIENTS WITH COMPUTER-ASSISTED
- 2: PATIENTS WITHOUT COMPUTER-ASSISTED

SUMMARY:
A poor outcome in anterior cruciate ligament (ACL) reconstruction is often related to tunnel position. The researchers believe that improving the accuracy of tunnel position will lead to an improved outcome in ACL surgery. The researchers' purpose is to perform a controlled study on a series of 500 patients in two groups: group I (250 cases) using conventional instrumentation and group II (250 cases) using navigation (Surgetics ACL Julliard protocol).

DETAILED DESCRIPTION:
This study compares the percentage of patients in 2 groups (full success) at 1 year of follow up. The results were evaluated on clinical outcome based on the IKDC (International Knee Documented Committee, subjective evaluation) form between one group using conventional instrumentation and another group using navigation.

Secondary Aims:

* To compare in 2 groups:

  * Gain of IKDC score at one year (based on pre-operative IKDC score)
  * Evolution of IKDC subjective (pre-operative, at 12 months)
* To compare performances at one year (% class A or B) in terms of initial instability measured with laximetry score
* Study of the learning curve
* Evaluate: lasting quality, complication rate, extra-operative time
* Evaluate frequency of thrombovenous complications
* Evaluate delay to return to sport

ELIGIBILITY:
Inclusion Criteria:

* First knee surgery
* Patients more than 18 years old

Exclusion Criteria:

* Knee surgery already done
* Patients unable to understand informed consent sheet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first knee surgery, available to control's visits at 6 months and one year
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2006-05; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
IKDC SCORE AT ONE YEAR | ONE YEAR

SECONDARY OUTCOMES:
COMPARISON IKDC SCORE BENEFIT AT ONE YEAR | one year
functionnal regaining between two groups at one year | one year
evaluate the surgeons' learning in the groups of patients with computer assisted | time of surgery, one year
evaluate hospitals' parameters in two groups | time of surgery, time of hospitalization
evaluate frequency of complication after surgery (infectious, thrombosis, scar) | 6 months, one year

CONTACTS AND LOCATIONS:
Overall Officials: Plaweski AP Stephane, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Beaufils P, Lerat JL. [Navigation for knee surgery]. Rev Chir Orthop Reparatrice Appar Mot. 2006 Sep;92(5 Suppl):2S199-2S207. No abstract available. French. PMID 17088785
- [Background] Plaweski S, Cazal J, Rosell P, Merloz P. Anterior cruciate ligament reconstruction using navigation: a comparative study on 60 patients. Am J Sports Med. 2006 Apr;34(4):542-52. doi: 10.1177/0363546505281799. PMID 16556753